CLINICAL TRIAL: NCT00048035
Title: An Open-label, Multicenter, Randomized Study to Determine Dose Conversion Factors at Different Frequencies of Administration After Switching From Maintenance Treatment With Intravenous Epoetin Alfa to Maintenance Treatment With Intravenous RO0503821 in Hemodialysis Patients With Chronic Renal Anemia.
Brief Title: A Study of Intravenous (iv) Mircera in Hemodialysis Patients With Chronic Renal Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16285
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (6):
- Cohort 1 (RO0503821 [0.25/150 1x/week]) (Experimental): Eligible participant will be administered RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) intravenously (IV) using a dose conversion factor of 0.25/150 microgram (mcg)/kilogram (kg) of the previous weekly erythropoiesis stimulating agents (ESA) dose, (equal to 62.50% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 2 (RO0503821 [0.25/150 1x/2week]) (Experimental): Eligible participant will be administered RO0503821 IV using a dose conversion factor of 0.25/150 mcg/kg of the previous weekly ESA dose, (equal to 62.50% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 3 (RO0503821 [0.4/150 1x/week]) (Experimental): Eligible participant will be administered RO0503821 IV using a dose conversion factor of 0.40/150 mcg/kg of the previous weekly ESA dose, (equal to100% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 4 (RO0503821 [0.4/150 1x/2week]) (Experimental): Eligible participant will be administered RO0503821 IV using a dose conversion factor of 0.40/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 5 (RO0503821 [0.6/150 1x/week]) (Experimental): Eligible participant will be administered RO0503821 IV using a dose conversion factor of 0.60/150 mcg/kg of the previous weekly ESA dose, (equal to150% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 6 (RO0503821 [0.6/150 1x/2week]) (Experimental): Eligible participant will be administered RO0503821 IV using a dose conversion factor of 0.60/150 mcg/kg of the previous weekly ESA dose, (equal to150% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — Differing doses and frequencies of iv administration

SUMMARY:
This study will determine the appropriate dose and frequency of administration of iv Mircera maintenance therapy in hemodialysis patients with chronic renal anemia who were previously receiving iv epoetin. The anticipated time on study treatment is 3-12 months and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* on hemodialysis therapy for at least 3 months;
* receiving iv epoetin alfa during the 2 weeks prior to the run-in period.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* use of any investigational drug within 30 days of the run-in phase, or during the run-in or study treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2002-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (13):
  - Birmingham, Alabama
  - Los Angeles, California
  - Maywood, Illinois
  - Louisville, Kentucky
  - Detroit, Michigan
  - Brooklyn Center, Minnesota
  - Las Vegas, Nevada
  - Paterson, New Jersey
  - Brooklyn, New York
  - Mineola, New York
  - New York, New York
  - Nashville, Tennessee
  - Morgantown, West Virginia

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 91 participants were enrolled in this study conducted from 19 March 2002 to 08 June 2005 at 14 Sites in United States.
Groups:
- Cohort 1 (RO0503821 [0.25/150 1x/ Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.25/150 mcg/kg of the previous weekly ESA dose, (equal to62.50% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 2 (RO0503821 [0.25/150 1x/2 Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.25/150 mcg/kg of the previous weekly ESA dose, (equal to62.50% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 3 (RO0503821 [0.4/150 1x/ Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.40/150 mcg/kg of the previous weekly ESA dose, (equal to100% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 4 (RO0503821 [0.4/150 1x/2week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.40/150 mcg/kg of the previous weekly ESA dose, (equal to100% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 5 (RO0503821 [0.6/150 1x/ Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.60/150 mcg/kg of the previous weekly ESA dose, (equal to150% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 6 (RO0503821 [0.6/150 1x/2 Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.60/150 mcg/kg of the previous weekly ESA dose, (equal to150% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1x/Week): Eligible participants were administered intravenously (IV) RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) once weekly (1x/ week) using a dose conversion factor of 0.25/150-, 0.40/150-, and 0.60/150 microgram (mcg)/kilogram (kg) of the previous weekly erythropoiesis stimulating agents (ESA) dose in Cohort 1, Cohort 3, and Cohort 5, respectively for 19 weeks. The ESA dose 62.5%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.25/150, 0.40/150 and 0.60/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1x/2Week): Eligible participants were administered IV RO0503821 once every two weeks (1x/ 2week) using a dose conversion factor of 0.25/150, 0.40/150, and 0.60/150 mcg/kg of the previous weekly ESA dose in Cohort 2, Cohort 4, and Cohort 6, respectively for 19 weeks. The ESA dose 62.5%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.25/150, 0.40/150 and 0.60/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
Period: Core Period
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/ Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2 Week]) | Cohort 3 (RO0503821 [0.4/150 1x/ Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/ Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2 Week]) | RO0503821 (1x/Week) | RO0503821 (1x/2Week)
Started | 15 | 15 | 15 | 15 | 16 | 15 | 0 | 0
Completed | 11 | 13 | 14 | 14 | 15 | 14 | 0 | 0
Not Completed | 4 | 2 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Early Withdrawals | 4 | 2 | 1 | 1 | 1 | 1 | 0 | 0
Period: Extension Year 1
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/ Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2 Week]) | Cohort 3 (RO0503821 [0.4/150 1x/ Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/ Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2 Week]) | RO0503821 (1x/Week) | RO0503821 (1x/2Week)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 27 (Participants (Cohorts 1, 3, and 5) who completed core, entered extension period (entry optional).) | 26 (Participants (Cohorts 2, 4 and 6) who completed core, entered extension period (entry optional).)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
Not completed — Early Withdrawals | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
Period: Extension Year 2
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/ Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2 Week]) | Cohort 3 (RO0503821 [0.4/150 1x/ Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/ Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2 Week]) | RO0503821 (1x/Week) | RO0503821 (1x/2Week)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 14 (A portion of participants who completed Extension Year 1, entered Extension Year 2 (entry optional).) | 13 (A portion of participants who completed Extension Year 1, entered Extension Year 2 (entry optional).)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Not completed — Early Withdrawals | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population was used for the analysis. It was defined as all randomized participants.
Groups:
- Cohort 1 (RO0503821 [0.25/150 1x/Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.25/150 mcg/kg of the previous weekly ESA dose, (equal to62.50% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 3 (RO0503821 [0.4/150 1x/Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.40/150 mcg/kg of the previous weekly ESA dose, (equal to100% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 5 (RO0503821 [0.6/150 1x/Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.60/150 mcg/kg of the previous weekly ESA dose, (equal to150% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2 Week]) | Cohort 3 (RO0503821 [0.4/150 1x/Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2 Week]) | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 16 | 15 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.90) | 58.6 (12.64) | 53.8 (12.72) | 62.8 (15.76) | 60.1 (11.89) | 62.5 (10.77) | 58.00 (12.91)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 8 | 6 | 6 | 6 | 3 | 31
  Male | 13 | 7 | 9 | 9 | 10 | 12 | 60

OUTCOME MEASURES:

1. Primary Outcome: Median Change From Baseline in Hemoglobin Levels to End of Initial Treatment Under Constant Dosing Regimen
Description: Median change from Baseline in hemoglobin (Hb) levels to end of initial treatment (EOIT) under constant dosing regimen was reported. For ease of interpretation, all individual slope values were multiplied by 42 to give an estimate of change in Hb values over six weeks. Baseline (Day -28 to Day 1) Hb values was calculated as the mean of the screening assessment (SA) and run-in period (Week -2 and Week -1). For all participants, an EOIT value was calculated as the last observed Hb value before a dose change or blood transfusion. For participants without any dose adjustments or blood transfusion, the EOIT value was identical to the Week 19 value.
Time Frame: From Baseline (Day -28 to Day 1) to EOIT (Week 19)
Population: The Intent-to-Treat (ITT) population was defined as all randomized participants.
Measure: Median (Inter-Quartile Range); unit: g/dL
Groups:
- Cohort 2 (RO0503821 [0.25/150 1x/2week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.25/150 mcg/kg of the previous weekly ESA dose, (equal to62.50% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 6 (RO0503821 [0.6/150 1x/2week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.60/150 mcg/kg of the previous weekly ESA dose, (equal to150% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2week]) | Cohort 3 (RO0503821 [0.4/150 1x/Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2week])
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 16 | 15
g/dL | -0.29 [-1.14 to 0.08] | -0.92 [-1.72 to 0.29] | -0.04 [-0.41 to 1.24] | -0.46 [-1.26 to -0.05] | 0.86 [0.15 to 1.31] | -0.07 [-0.93 to 0.48]
Statistical Analysis 1: Comparison: Cohort 1 (RO0503821 [0.25/150 1x/Week]) vs Cohort 3 (RO0503821 [0.4/150 1x/Week]) vs Cohort 5 (RO0503821 [0.6/150 1x/Week]); All cohorts with dosing frequency 1 X / Week; Test type: Superiority or Other; Estimated Conversion Factor 90% CI = 0.38, 90% CI 2-sided [0.32 to 0.42] — To analyze the appropriateness of the chosen dose conversion factors, a second regression analysis was carried out. This was a regression on the three different conversion factor dose groups, using the regression slope estimates of Hb
Statistical Analysis 2: Comparison: Cohort 2 (RO0503821 [0.25/150 1x/2week]) vs Cohort 4 (RO0503821 [0.4/150 1x/2week]) vs Cohort 6 (RO0503821 [0.6/150 1x/2week]); All cohorts with dosing frequency 1 X /2 Week; Test type: Superiority or Other; Estimated Conversion Factor 90% CI = 0.61, 90% CI 2-sided [0.53 to 0.76] — To analyze the appropriateness of the chosen dose conversion factors, a second regression analysis was carried out. This was a regression on the three different conversion factor dose groups, using the regression slope estimates of Hb change

2. Secondary Outcome: Median Change From Baseline in Hematocrit Levels to End of Initial Treatment Under Constant Dosing Regimen
Description: Median change from Baseline in hematocrit (Hct) levels to end of initial treatment under constant dosing regimen was reported. Baseline (Day -28 to Day 1) Hct values was calculated as the mean of the SA and run-in period (Weeks -2 and -1). For all participants, an EOIT value was calculated as the last observed Hct value before a dose change or blood transfusion. For participants without any dose adjustments or blood transfusion, the EOIT value was identical to the Week 19 value.
Time Frame: From Baseline (Day -28 to Day 1) to EOIT (Week 19)
Population: The Intent-to-Treat (ITT) population was defined as all randomized participants.
Measure: Median (Inter-Quartile Range); unit: g/dL
Groups:
- Cohort 1 (RO0503821 [0.25/150 1x/Week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.25/150 mcg/kg of the previous weekly ESA dose, (equal to 62.50% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 2 (RO0503821 [0.25/150 1x/2week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.25/150 mcg/kg of the previous weekly ESA dose, (equal to 62.50% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort 4 (RO0503821 [0.4/150 1x/2week]): Eligible participant were administered RO0503821 IV using a dose conversion factor of 0.40/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once in every two weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2week]) | Cohort 3 (RO0503821 [0.4/150 1x/Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2week])
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 16 | 15
g/dL | -1.50 [-3.31 to 0.30] | -3.01 [-5.14 to -0.89] | -0.32 [-1.26 to 4.08] | -1.62 [-4.25 to -0.21] | 2.73 [0.37 to 4.28] | -0.07 [-2.57 to 1.51]

3. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Events, And Deaths
Description: An Adverse Events (AEs) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious Adverse Events (SAEs) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes. ). The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time all results for the two long term safety periods were displayed by dose schedule group only.
Time Frame: Up to Week 126
Population: The safety population was considered for analysis which included all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- RO0503821 (1x/Week): Eligible participants were administered IV RO0503821 once weekly (1x/ week) using a dose conversion factor of 0.25/150, 0.40/150, and 0.60/150 mcg/kg of the previous weekly ESA dose in Cohort 1, Cohort 3, and Cohort 5, respectively for 19 weeks. The ESA dose 62.5%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.25/150, 0.40/150 and 0.60/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
Arm/Group | RO0503821 (1x/Week) | RO0503821 (1x/2Week)
Number analyzed (Participants) | 46 | 45
Participants
  Any AEs | 42 | 37
  Any SAEs | 20 | 20
  Deaths | 3 | 2

4. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Marked abnormality was defined as above and/or below a value which was considered to be potentially clinically relevant. The number of participants with marked lab abnormality across treatment groups were reported and presented. Marked laboratory abnormalities were analyzed according to the Roche specified limits for the following reference range: White blood cells (WBC) (3.0- 18.0 10^9/L), Platelets (100 - 550 10^9/L), Alanine aminotransferase (ALAT) [0 110 units per litre (U/L)], Alkaline Phosphatase (ALP) (0 - 220 U/L), Aspartate aminotransferase (ASAT) (0 - 80 U/L), Albumin >= 30 g/L, Phosphate [0.75 - 1.60 millimoles per liter (mmol/L)], Potassium (2.9 - 5.8 mmol/L), Glucose (2.80 - 11.10 mmol/L).
Time Frame: Up to Week 126
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2week]) | Cohort 3 (RO0503821 [0.4/150 1x/Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2week])
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 16 | 15
Participants
  Phosphate -High; (n = 15, 15, 15, 15 , 16 , 15) | 3 | 1 | 3 | 4 | 4 | 2
  Phosphate -Low; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 1 | 1 | 0 | 2 | 0
  Potassium -High; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 1 | 0 | 2 | 0
  Potassium -Low; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  Platelets - High; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  Platelets - Low; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 1 | 1 | 0 | 0
  WBC - High; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  WBC - Low; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 1 | 1 | 0 | 0
  Basophils - High; (n = 15, 15, 14, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils - High; (n = 15, 15, 14, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes - High; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes - Low; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 3 | 2 | 1 | 2 | 3
  Monocytes - High; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes - Low; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils - Low; (n = 15, 15, 14, 15 , 16 , 15) | 0 | 0 | 0 | 1 | 0 | 0
  ALAT - High; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 1 | 0 | 0 | 0
  ALP - High; (n = 15, 15, 15, 15 , 16 , 15) | 1 | 0 | 1 | 0 | 0 | 1
  ASAT - High; (n = 15, 15, 15, 15 , 16 , 15) | 0 | 0 | 1 | 0 | 0 | 0
  Total Bilirubin-High; (n = 15, 15, 15, 15, 16, 15) | 0 | 0 | 0 | 0 | 0 | 1
  Albumin - Low; (n = 15, 15, 15, 15 , 16 , 15) | 1 | 0 | 0 | 0 | 0 | 0
  Glucose Fasting -High; (n = 5, 6, 9, 6, 6 , 9) | 0 | 0 | 0 | 0 | 0 | 0
  Glucose Fasting -Low; (n = 5, 6, 9, 6, 6 , 9) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure Before and After Dialysis
Description: Mean Change from Baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) is calculated as the end of treatment values minus the Baseline value. Baseline (Day -28 to Day 1) values were calculated as the mean of the screening assessment (SA) and run-in period (Week -2 and Week -1).
Time Frame: From Baseline (Day -28 to Day 1) to Week 126
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2week]) | Cohort 3 (RO0503821 [0.4/150 1x/Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2week])
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 16 | 15
mm HG
  DBP- before dialysis | -2 (12.2) | -1 (14.7) | -10 (12.4) | -8 (14.3) | -6 (13.1) | -10 (12.4)
  DBP - After dialysis | 4 (16.7) | 0 (19.0) | -0 (14.5) | -8 (18.0) | -6 (18.1) | -0 (14.5)
  SBP - before dialysis | -1 (26.4) | 5 (25.5) | -15 (21.6) | -15 (23.8) | -11 (21.7) | -15 (21.6)
  SBP - After dialysis | 6 (30.1) | 3 (26.5) | -3 (30.4) | -13 (26.7) | -6 (27.1) | -3 (30.4)

6. Secondary Outcome: Mean Change in Pulse Rate
Description: Participants pulse rates in beats per minute (BpM) were analyzed at sitting position using descriptive statistical methods (ie, means, standard deviations and percentiles). The changes in pulse rate throughout the study were analysed at each study visit and mean change is reported.
Time Frame: Up to Week 126
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: BpM
Arm/Group | Cohort 1 (RO0503821 [0.25/150 1x/Week]) | Cohort 2 (RO0503821 [0.25/150 1x/2week]) | Cohort 3 (RO0503821 [0.4/150 1x/Week]) | Cohort 4 (RO0503821 [0.4/150 1x/2week]) | Cohort 5 (RO0503821 [0.6/150 1x/Week]) | Cohort 6 (RO0503821 [0.6/150 1x/2week])
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 16 | 15
BpM | -1 (10.1) | 1 (14.8) | 2 (10.5) | 3 (14.1) | -1 (10.2) | 3 (12.6)

ADVERSE EVENTS:
Time Frame: Up to Week 126
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis population. The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time all results for the two long term safety periods were displayed by dose schedule group only.
Groups:
- RO0503821 (1/Week): Eligible participants were administered IV RO0503821 once weekly (1x/ week) using a dose conversion factor of 0.25/150, 0.40/150, and 0.60/150 mcg/kg of the previous weekly ESA dose in Cohort 1, Cohort 3, and Cohort 5, respectively for 19 weeks. The ESA dose 62.5%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.25/150, 0.40/150 and 0.60/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1/2week): Eligible participants were administered IV RO0503821 once every two weeks (1x/ 2week) using a dose conversion factor of 0.25/150-, 0.40/150-, and 0.60/150 mcg/kg of the previous weekly ESA dose in Cohort 2, Cohort 4, and Cohort 6, respectively for 19 weeks. The ESA dose 62.5%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.25/150, 0.40/150 and 0.60/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
Arm/Group | RO0503821 (1/Week) | RO0503821 (1/2week)
Serious Adverse Events (participants affected / at risk) | 20/46 | 20/45
Other Adverse Events (participants affected / at risk) | 34/46 | 30/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1/Week) (N=46) | RO0503821 (1/2week) (N=45)
Cardiac Failure Congestive (Cardiac disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Ischaemic ulcer (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Ileostomy closure (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1/Week) (N=46) | RO0503821 (1/2week) (N=45)
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Gastritis (Gastrointestinal disorders) | 0 | 3
Vascular access complication (Injury, poisoning and procedural complications) | 5 | 4
Procedural hypotension (Injury, poisoning and procedural complications) | 3 | 5
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 6 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3 | 2
Fatigue (General disorders) | 5 | 6
Pyrexia (General disorders) | 3 | 7
Chest pain (General disorders) | 3 | 5
Asthenia (General disorders) | 0 | 4
Chest discomfort (General disorders) | 1 | 3
Headache (Nervous system disorders) | 10 | 4
Dizziness (Nervous system disorders) | 4 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 0
Hypertension (Vascular disorders) | 3 | 3
Cataract (Eye disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.